CLINICAL TRIAL: NCT01720446
Title: A Long-term, Randomised, Double-blind, Placebo-controlled, Multinational, Multi-centre Trial to Evaluate Cardiovascular and Other Long-term Outcomes With Semaglutide in Subjects With Type 2 Diabetes (SUSTAIN™ 6 - Long-term Outcomes)
Brief Title: Trial to Evaluate Cardiovascular and Other Long-term Outcomes With Semaglutide in Subjects With Type 2 Diabetes
Acronym: SUSTAIN™ 6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3744; 2012-002839-28 (EudraCT Number); U1111-1131-7227 (Other: WHO)
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Results first posted 2018-03-15 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Semaglutide 0.5 mg (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide 1.0 mg (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide placebo 0.5 mg (Placebo Comparator)
  Interventions: Drug: placebo
- Semaglutide placebo 1.0 mg (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Once weekly doses of 0.5 mg semaglutide after an initial dose escalation step of 0.25 mg as an add-on to the standard-of-care treatment. Administered subcutaneously (s.c., under the skin)
  Arms: Semaglutide 0.5 mg
Drug: semaglutide — Once weekly doses of 1.0 mg semaglutide after an initial dose escalation step of 0.25 mg followed by 0.5 mg dose escalation as an add-on to the standard-of-care treatment. Administered subcutaneously (s.c., under the skin)
  Arms: Semaglutide 1.0 mg
Drug: placebo — Once weekly doses volume-matched placebo, as an add-on to the standard-of-care treatment. Administered subcutaneously (s.c., under the skin).
  Arms: Semaglutide placebo 0.5 mg; Semaglutide placebo 1.0 mg

SUMMARY:
This trial is conducted globally. The aim of the trial is to evaluate cardiovascular and other long-term outcomes with semaglutide in subjects with type 2 diabetes. The trial is event-driven, i.e. the maximum trial duration (up to max. 148 weeks) will depend on the accrual of major adverse cardiovascular events (MACE) in this trial and the remaining research programme. The incidence of MACE will be monitored throughout the trial which will be terminated according to plan when pre-specified stopping criteria are met.

ELIGIBILITY:
Inclusion Criteria: - Men and women with type 2 diabetes mellitus - Age above or equal to 50 years at screening and clinical evidence of cardiovascular disease or age above or equal to 60 years at screening and subclinical evidence of cardiovascular disease - Anti-diabetic drug naïve, or treated with one or two oral antidiabetic drug (OADs), or treated with human Neutral Protamin Hagedorn (NPH) insulin or long-acting insulin analogue or pre-mixed insulin, both types of insulin either alone or in combination with one or two OADs - HbA1c above or equal to 7.0% at screening Exclusion Criteria: - Type 1 diabetes mellitus - Use of glucagon-like peptide-1 (GLP-1) receptor agonist (exenatide, liraglutide, or other) or pramlintide within 90 days prior to screening - Use of any dipeptidyl peptidase 4 (DPP-IV) inhibitor within 30 days prior to screening - Treatment with insulin other than basal and pre-mixed insulin within 90 days prior to screening - except for short-term use in connection with intercurrent illness - Acute decompensation of glycaemic control requiring immediate intensification of treatment to prevent acute complications of diabetes (eg diabetes ketoacidosis) within 90 days prior to screening - History of chronic pancreatitis or idiopathic acute pancreatitis - Acute coronary or cerebro-vascular event within 90 days prior to randomisation - Currently planned coronary, carotid or peripheral artery revascularisation - Chronic heart failure New York Heart Association (NYHA) class IV - Personal or family history of multiple endocrine neoplasia type 2 (MEN2) or familial medullary thyroid carcinoma - Personal history of non-familial medullary thyroid carcinoma - Screening calcitonin above or equal to 50 ng/L

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3297 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (218):
- United States (87):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Chandler, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Crystal River, Florida
  - Novo Nordisk Investigational Site, DeLand, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Ponte Vedra, Florida
  - Novo Nordisk Investigational Site, Spring Hill, Florida
  - Novo Nordisk Investigational Site, St. Petersburg, Florida
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Michigan City, Indiana
  - Novo Nordisk Investigational Site, Mishawaka, Indiana
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Monroe, Louisiana
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Methuen, Massachusetts
  - Novo Nordisk Investigational Site, North Dartmouth, Massachusetts
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Lebanon, New Hampshire
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Mine Hill, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, McMurray, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Bartlett, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Longview, Texas
  - Novo Nordisk Investigational Site, Odessa, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, South Burlington, Vermont
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Wenatchee, Washington
  - Novo Nordisk Investigational Site, Madison, Wisconsin
- Algeria (4):
  - Novo Nordisk Investigational Site, Annaba
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Sétif
  - Novo Nordisk Investigational Site, Tizi Ouzou
- Argentina (4):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Mar del Plata
  - Novo Nordisk Investigational Site, Morón
- Australia (8):
  - Novo Nordisk Investigational Site, Blacktown, New South Wales
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Ipswich, Queensland
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, Oaklands Park, South Australia
  - Novo Nordisk Investigational Site, Box Hill, Victoria
  - Novo Nordisk Investigational Site, Fitzroy, Victoria
  - Novo Nordisk Investigational Site, Fremantle, Western Australia
- Brazil (5):
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Belém, Pará
  - Novo Nordisk Investigational Site, Campinas, São Paulo
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Porto Alegre
- Bulgaria (3):
  - Novo Nordisk Investigational Site, Pleven
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Canada (14):
  - Novo Nordisk Investigational Site, Calgary, Alberta
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Cambridge, Ontario
  - Novo Nordisk Investigational Site, Cornwall, Ontario
  - Novo Nordisk Investigational Site, London, Ontario
  - Novo Nordisk Investigational Site, Smiths Falls, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Waterloo, Ontario
  - Novo Nordisk Investigational Site, Drummondville, Quebec
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Victoriaville, Quebec
  - Novo Nordisk Investigational Site, Québec
- Denmark (5):
  - Novo Nordisk Investigational Site, Aarhus C
  - Novo Nordisk Investigational Site, Gentofte Municipality
  - Novo Nordisk Investigational Site, Hellerup
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Odense
- Germany (8):
  - Novo Nordisk Investigational Site, Elsterwerda
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Freiburg im Breisgau
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Oldenburg
  - Novo Nordisk Investigational Site, Saint Ingbert
- India (14):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Visakhapatnam, Andhra Pradesh
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Mysore, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Delhi, New Delhi
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
  - Novo Nordisk Investigational Site, Pune
- Israel (6):
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Nahariya
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Tel Litwinsky
- Italy (6):
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Olbia
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Primo Piano Palazzina Ambulato
  - Novo Nordisk Investigational Site, Siena
- Malaysia (6):
  - Novo Nordisk Investigational Site, Kota Samarahan
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Kuching
  - Novo Nordisk Investigational Site, Malacca
  - Novo Nordisk Investigational Site, Serdang
  - Novo Nordisk Investigational Site, Seremban
- Mexico (7):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Cuernavaca, Morelos
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, México D.F., México, D.F.
  - Novo Nordisk Investigational Site, Ciudad Madero, Tamaulipas
  - Novo Nordisk Investigational Site, Aguascalientes
  - Novo Nordisk Investigational Site, San Luis Potosí City
- Poland (5):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zabrze
- Russia (10):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Smolensk
  - Novo Nordisk Investigational Site, Yaroslavl
- Spain (6):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Antequera
  - Novo Nordisk Investigational Site, Pozuelo de Alarcón
  - Novo Nordisk Investigational Site, Sanlúcar de Barrameda - Cádiz-
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Vic (Barcelona)
- Taiwan (4):
  - Novo Nordisk Investigational Site, Chiayi City
  - Novo Nordisk Investigational Site, Tainan
  - Novo Nordisk Investigational Site, Taipei
  - Novo Nordisk Investigational Site, Taoyuan District
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (7):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Çanakkale
  - Novo Nordisk Investigational Site, Denizli
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Kocaeli
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, Northwood
  - Novo Nordisk Investigational Site, Sidcup
  - Novo Nordisk Investigational Site, Swansea
  - Novo Nordisk Investigational Site, Torquay

REFERENCES:
- [Background] Verma S, Bain SC, Monk Fries T, Mazer CD, Nauck MA, Pratley RE, Rasmussen S, Saevereid HA, Zinman B, Buse JB. Duration of diabetes and cardiorenal efficacy of liraglutide and semaglutide: A post hoc analysis of the LEADER and SUSTAIN 6 clinical trials. Diabetes Obes Metab. 2019 Jul;21(7):1745-1751. doi: 10.1111/dom.13698. Epub 2019 Apr 2. PMID 30851070
- [Result] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Result] Vilsboll T, Bain SC, Leiter LA, Lingvay I, Matthews D, Simo R, Helmark IC, Wijayasinghe N, Larsen M. Semaglutide, reduction in glycated haemoglobin and the risk of diabetic retinopathy. Diabetes Obes Metab. 2018 Apr;20(4):889-897. doi: 10.1111/dom.13172. Epub 2018 Jan 8. PMID 29178519
- [Result] Carlsson Petri KC, Ingwersen SH, Flint A, Zacho J, Overgaard RV. Semaglutide s.c. Once-Weekly in Type 2 Diabetes: A Population Pharmacokinetic Analysis. Diabetes Ther. 2018 Aug;9(4):1533-1547. doi: 10.1007/s13300-018-0458-5. Epub 2018 Jun 15. PMID 29907893
- [Result] Aroda VR, Ahmann A, Cariou B, Chow F, Davies MJ, Jodar E, Mehta R, Woo V, Lingvay I. Comparative efficacy, safety, and cardiovascular outcomes with once-weekly subcutaneous semaglutide in the treatment of type 2 diabetes: Insights from the SUSTAIN 1-7 trials. Diabetes Metab. 2019 Oct;45(5):409-418. doi: 10.1016/j.diabet.2018.12.001. Epub 2019 Jan 4. PMID 30615985
- [Result] Leiter LA, Bain SC, Hramiak I, Jodar E, Madsbad S, Gondolf T, Hansen T, Holst I, Lingvay I. Cardiovascular risk reduction with once-weekly semaglutide in subjects with type 2 diabetes: a post hoc analysis of gender, age, and baseline CV risk profile in the SUSTAIN 6 trial. Cardiovasc Diabetol. 2019 Jun 6;18(1):73. doi: 10.1186/s12933-019-0871-8. PMID 31167654
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Bain SC, Belmar N, Hoff ST, Husain M, Rasmussen S, Vilsboll T, Petrie MC. Cardiovascular, Metabolic, and Safety Outcomes with Semaglutide by Baseline Age: Post Hoc Analysis of SUSTAIN 6 and PIONEER 6. Diabetes Ther. 2025 Jan;16(1):15-28. doi: 10.1007/s13300-024-01659-7. Epub 2024 Nov 9. PMID 39520501
- [Derived] Rossing P, Bain SC, Bosch-Traberg H, Sokareva E, Heerspink HJL, Rasmussen S, Mellbin LG. Effect of semaglutide on major adverse cardiovascular events by baseline kidney parameters in participants with type 2 diabetes and at high risk of cardiovascular disease: SUSTAIN 6 and PIONEER 6 post hoc pooled analysis. Cardiovasc Diabetol. 2023 Aug 24;22(1):220. doi: 10.1186/s12933-023-01949-7. PMID 37620807
- [Derived] Strain WD, Frenkel O, James MA, Leiter LA, Rasmussen S, Rothwell PM, Sejersten Ripa M, Truelsen TC, Husain M. Effects of Semaglutide on Stroke Subtypes in Type 2 Diabetes: Post Hoc Analysis of the Randomized SUSTAIN 6 and PIONEER 6. Stroke. 2022 Sep;53(9):2749-2757. doi: 10.1161/STROKEAHA.121.037775. Epub 2022 May 18. PMID 35582947
- [Derived] Husain M, Consoli A, De Remigis A, Pettersson Meyer AS, Rasmussen S, Bain S. Semaglutide reduces cardiovascular events regardless of metformin use: a post hoc subgroup analysis of SUSTAIN 6 and PIONEER 6. Cardiovasc Diabetol. 2022 Apr 28;21(1):64. doi: 10.1186/s12933-022-01489-6. PMID 35484580
- [Derived] Verma S, Al-Omran M, Leiter LA, Mazer CD, Rasmussen S, Saevereid HA, Sejersten Ripa M, Bonaca MP. Cardiovascular efficacy of liraglutide and semaglutide in individuals with diabetes and peripheral artery disease. Diabetes Obes Metab. 2022 Jul;24(7):1288-1299. doi: 10.1111/dom.14700. Epub 2022 Apr 11. PMID 35332654
- [Derived] Verma S, Fainberg U, Husain M, Rasmussen S, Ryden L, Ripa MS, Buse JB. Applying REWIND cardiovascular disease criteria to SUSTAIN 6 and PIONEER 6: An exploratory analysis of cardiovascular outcomes with semaglutide. Diabetes Obes Metab. 2021 Jul;23(7):1677-1680. doi: 10.1111/dom.14360. Epub 2021 Mar 18. PMID 33606902
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Verma S, McGuire DK, Bain SC, Bhatt DL, Leiter LA, Mazer CD, Monk Fries T, Pratley RE, Rasmussen S, Vrazic H, Zinman B, Buse JB. Effects of glucagon-like peptide-1 receptor agonists liraglutide and semaglutide on cardiovascular and renal outcomes across body mass index categories in type 2 diabetes: Results of the LEADER and SUSTAIN 6 trials. Diabetes Obes Metab. 2020 Dec;22(12):2487-2492. doi: 10.1111/dom.14160. Epub 2020 Sep 4. PMID 32744418
- [Derived] Verma S, Bain SC, Honore JB, F E Mann J, A Nauck M, E Pratley R, Rasmussen S, Sejersten Ripa M, Zinman B, Buse JB. Impact of microvascular disease on cardiovascular outcomes in type 2 diabetes: Results from the LEADER and SUSTAIN 6 clinical trials. Diabetes Obes Metab. 2020 Nov;22(11):2193-2198. doi: 10.1111/dom.14140. Epub 2020 Aug 12. PMID 32643857
- [Derived] Leiter LA, Bain SC, Bhatt DL, Buse JB, Mazer CD, Pratley RE, Rasmussen S, Ripa MS, Vrazic H, Verma S. The effect of glucagon-like peptide-1 receptor agonists liraglutide and semaglutide on cardiovascular and renal outcomes across baseline blood pressure categories: Analysis of the LEADER and SUSTAIN 6 trials. Diabetes Obes Metab. 2020 Sep;22(9):1690-1695. doi: 10.1111/dom.14079. Epub 2020 Jun 3. PMID 32372454
- [Derived] Jodar E, Michelsen M, Polonsky W, Rea R, Sandberg A, Vilsboll T, Warren M, Harring S, Ziegler U, Bain S. Semaglutide improves health-related quality of life versus placebo when added to standard of care in patients with type 2 diabetes at high cardiovascular risk (SUSTAIN 6). Diabetes Obes Metab. 2020 Aug;22(8):1339-1347. doi: 10.1111/dom.14039. Epub 2020 Apr 27. PMID 32227613
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- [Derived] DeSouza C, Cariou B, Garg S, Lausvig N, Navarria A, Fonseca V. Efficacy and Safety of Semaglutide for Type 2 Diabetes by Race and Ethnicity: A Post Hoc Analysis of the SUSTAIN Trials. J Clin Endocrinol Metab. 2020 Feb 1;105(2):dgz072. doi: 10.1210/clinem/dgz072. PMID 31769496
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Generalizability of glucagon-like peptide-1 receptor agonist cardiovascular outcome trials enrollment criteria to the US type 2 diabetes population. Am J Manag Care. 2018 Apr;24(8 Suppl):S146-S155. PMID 29693361
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 229 sites in 20 countries. Country (sites): Algeria (4), Argentina (7), Australia (8), Brazil (8), Bulgaria (5), Canada (13), Denmark (5), Germany (7), Israel (6), Italy (6), Malaysia (6), Mexico (9), Poland (5), Russia (11), Spain (6), Taiwan (4), Thailand (5), Turkey (10), United Kingdom (8) and United States (96).
Pre-assignment Details: Subjects could be anti-glycaemic drug naïve, or treated with 1 or 2 oral anti diabetic drugs (OADs), or treated with human NPH insulin or long-acting insulin analogue or pre-mixed insulin, alone or in combination with 1 or 2 OAD(s).
Groups:
- Semaglutide 0.5 mg: Subjects received once-weekly dose of semaglutide 0.5 mg as an add-on to their standard-of-care treatment. Injections were administered subcutaneously in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same weekday during the trial. Semaglutide was initiated at a dose of 0.25 mg and was escalated (doubled) to 0.5 mg after 4 weeks. Hence the target dose of 0.5 mg was achieved after 4 weeks of treatment. Each subject was treated for 104 weeks.
- Semaglutide 1.0 mg: Subjects received once-weekly dose of semaglutide 1.0 mg as an add-on to their standard-of-care treatment. Injections were administered subcutaneously in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same weekday during the trial. Semaglutide was initiated at a dose of 0.25 mg and was escalated (doubled) to 0.5 mg after 4 weeks. Hence the target dose of 1.0 mg was achieved after 8 weeks of treatment. Each subject was treated for 104 weeks.
- Placebo 0.5 mg: Subjects received once-weekly dose of placebo 0.5 mg as an add-on to their standard-of-care treatment. Injections were administered subcutaneously in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same weekday during the trial. Placebo was initiated at a dose of 0.25 mg and was escalated (doubled) to 0.5 mg after 4 weeks. Hence the target dose of 0.5 mg was achieved after 4 weeks of treatment. Each subject was treated for 104 weeks.
- Placebo 1.0 mg: Subjects received once-weekly dose of placebo 1.0 mg as an add-on to their standard-of-care treatment. Injections were administered subcutaneously in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same weekday during the trial. Placebo was initiated at a dose of 0.25 mg and was escalated (doubled) to 0.5 mg after 4 weeks. Hence the target dose of 1.0 mg was achieved after 8 weeks of treatment. Each subject was treated for 104 weeks.
Period: Overall Study
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Started | 826 | 822 | 824 | 825
Premature Treatment Discontinuers | 164 (Premature treatment discontinuers were allowed to continue participation in the trial.) | 186 (Premature treatment discontinuers were allowed to continue participation in the trial.) | 151 (Premature treatment discontinuers were allowed to continue participation in the trial.) | 159 (Premature treatment discontinuers were allowed to continue participation in the trial.)
Completed | 812 (Subjects who did not permanently discontinue treatment prematurely.) | 811 (Subjects who did not permanently discontinue treatment prematurely.) | 804 (Subjects who did not permanently discontinue treatment prematurely.) | 805 (Subjects who did not permanently discontinue treatment prematurely.)
Not Completed | 14 | 11 | 20 | 20
Not completed — Lost to Follow-up | 12 | 6 | 16 | 16
Not completed — Withdrawal by Subject | 2 | 5 | 4 | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on full analysis set which included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg | Total
Number analyzed (Participants) | 826 | 822 | 824 | 825 | 3297
Age, Customized [Number; unit: participants]
  50-64 years | 440 | 415 | 419 | 425 | 1699
  65-74 years | 312 | 324 | 324 | 317 | 1277
  75-84 years | 71 | 76 | 75 | 79 | 301
  85 and over | 3 | 7 | 6 | 4 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 331 | 304 | 342 | 318 | 1295
  Male | 495 | 518 | 482 | 507 | 2002
Glycosylated haemoglobin [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.67 (1.39) | 8.73 (1.51) | 8.70 (1.49) | 8.70 (1.45) | 8.70 (1.46)
Fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] | 185.4 (66.09) | 182.9 (68.04) | 185.8 (68.23) | 184.6 (63.08) | 184.7 (66.37)
Body weight [Mean (Standard Deviation); unit: kg] | 91.80 (20.25) | 92.86 (21.05) | 91.83 (20.35) | 91.90 (20.75) | 92.09 (20.60)
LDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 89.62 (39.08) | 89.72 (34.49) | 89.01 (38.35) | 91.14 (37.90) | 89.87 (37.49)
HDL-cholesterol [Mean (Standard Deviation); unit: mg/dL] | 45.92 (13.00) | 44.97 (12.42) | 45.82 (12.92) | 44.61 (12.26) | 45.33 (12.66)
Systolic BP [Mean (Standard Deviation); unit: mmHg] | 136.1 (17.97) | 135.8 (16.96) | 135.8 (16.16) | 134.8 (17.45) | 135.6 (17.15)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 77.10 (9.78) | 76.88 (10.21) | 77.54 (9.85) | 76.66 (10.21) | 77.05 (10.02)
Pulse rate [Mean (Standard Deviation); unit: beats/min] | 72.69 (11.22) | 71.53 (10.86) | 72.01 (10.62) | 71.95 (10.92) | 72.05 (10.91)
Total cholesterol [Geometric Mean (Full Range); unit: mg/dL] | 165.38 [65.25 to 632.43] | 164.96 [79.54 to 562.16] | 164.38 [70.27 to 378.38] | 165.97 [64.86 to 537.07] | 165.17 [64.86 to 632.43]
Triglycerides [Geometric Mean (Full Range); unit: mg/dL] | 163.66 [27.59 to 1913.50] | 158.93 [10.68 to 3378.44] | 162.30 [30.26 to 1438.24] | 163.00 [35.60 to 2435.93] | 161.96 [10.68 to 3378.44]
Free fatty acids [Geometric Mean (Full Range); unit: mmol/L] | 0.83 [0.04 to 3.82] | 0.80 [0.04 to 4.20] | 0.83 [0.04 to 3.34] | 0.81 [0.04 to 4.22] | 0.82 [0.04 to 4.22]

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomisation to First Occurrence of a MACE, Defined as Cardiovascular Death, Non-fatal Myocardial Infarction, or Non-fatal Stroke
Description: Percentage of subjects experiencing a first event of a major adverse cardiovascular event (MACE), defined as cardiovascular (CV) death, non-fatal myocardial infarction (MI), or non-fatal stroke.
Time Frame: Time from randomisation up to end of follow-up (scheduled at week 109)
Population: Full analysis set included all the randomised subjects. As specified in the protocol, the two semaglutide dose arms (semaglutide 0.5 mg + semaglutide 1.0 mg) and the two placebo dose arms (placebo 0.5 mg + placebo 1.0 mg) were pooled for the analysis of this endpoint.
Measure: Number; unit: percentage of subjects
Groups:
- Semaglutide: Subjects received once-weekly dose of semaglutide 0.5 mg or 1.0 mg as an add-on to their standard-of-care treatment. Injections were administered subcutaneously in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same weekday during the trial. Semaglutide was initiated at a dose of 0.25 mg and was escalated (doubled) to 0.5 mg after 4 weeks. Hence the target dose of 0.5 mg was achieved after 4 weeks of treatment and the target dose of 1.0 mg was achieved after 8 weeks of treatment. Each subject was treated for 104 weeks.
- Placebo: Subjects received once-weekly dose of placebo 0.5 mg or 1.0 mg as an add-on to their standard-of-care treatment. Injections were administered subcutaneously in the thigh, abdomen or upper arm, at any time of day irrespective of meals. The injections were to be administered on the same weekday during the trial. Placebo was initiated at a dose of 0.25 mg and was escalated (doubled) to 0.5 mg after 4 weeks. Hence the target dose of 0.5 mg was achieved after 4 weeks of treatment and the target dose of 1.0 mg was achieved after 8 weeks of treatment. Each subject was treated for 104 weeks.
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1648 | 1649
percentage of subjects | 6.6 | 8.9
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; The primary endpoint was analysed using a stratified Cox proportional hazards model with treatment group (semaglutide, placebo) as fixed factor. Assuming the same population MACE risk for the semaglutide and placebo groups (i.e., the population hazards ratio [HR] equals 1), a total minimum of 122 events were needed in order to have at least 90% power to ascertain that the upper two-sided 95% confidence limit for the HR was less than 1.8; Test type: Non-Inferiority or Equivalence — Non-inferiority of semaglutide versus placebo was considered to be confirmed if the upper limit of the two-sided 95% CI for the HR was below 1.8 or equivalent if the p-value for the one-sided test of: H0: HR ≥ 1.8 against Ha: HR <1.8 was less than 2.5% (or equivalent to 5% for a two-sided test); p < 0.0001, Regression, Cox — The 'p-value' is for the two-sided Wald test of non-inferiority with limit 1.8; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.58 to 0.95] — Semaglutide/Placebo
Statistical Analysis 2: Comparison: Semaglutide vs Placebo; A post hoc analysis of superiority of semaglutide versus placebo was performed based on the pre-specified Cox proportional hazard analysis using the two-sided Wald test of no difference, with treatment (semaglutide, placebo) as fixed factor and stratified by all possible combinations of the three stratification factors used in the randomisation procedure (in total 9 levels); Test type: Superiority or Other; p = 0.0167, Regression, Cox — The 'p-value' is for the two-sided Wald test of no difference; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.58 to 0.95] — Semaglutide/Placebo

2. Secondary Outcome: Time From Randomisation to First Occurrence of an Expanded Composite Cardiovascular Outcome
Description: Percentage of subjects experiencing first occurrence of an expanded composite CV outcome (defined as either MACE, revascularisation [coronary and peripheral], unstable angina requiring hospitalisation or hospitalisation for heart failure)
Time Frame: Time from randomisation up to end of follow-up (scheduled at week 109)
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1648 | 1649
percentage of subjects | 12.1 | 16.0
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Analysis was done by Cox proportional hazards model with treatment (semaglutide; placebo) as a fixed factor and stratified by all possible combinations of the three stratification factors used in the randomisation procedure (in total 9 levels); Test type: Superiority or Other; p = 0.0016, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.62 to 0.89] — Semaglutide/Placebo

3. Secondary Outcome: Time From Randomisation to Each Individual Component of the Expanded Composite Cardiovascular Outcome
Description: Percentage of subjects experiencing an event onset for each individual component of the expanded composite cardiovascular outcomes (defined as either MACE, revascularisation [coronary and peripheral], unstable angina requiring hospitalisation or hospitalisation for heart failure).
Time Frame: Time from randomisation up to end of follow-up (scheduled at week 109)
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1648 | 1649
percentage of subjects
  Cardiovascular death | 1.6 | 1.9
  Non-fatal MI | 2.5 | 3.7
  Non-fatal Stroke | 1.5 | 2.5
  Revascularisation | 2.6 | 4.2
  UAP requiring hospitalisation | 1.1 | 1.3
  Hospitalisation for heart failure | 2.7 | 2.4
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Analysis for CV death was done by Cox proportional hazards model with treatment (semaglutide; placebo) as a fixed factor and stratified by all possible combinations of the three stratification factors used in the randomisation procedure (in total 9 levels); Test type: Superiority or Other; p = 0.9181, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.65 to 1.48] — Semaglutide/Placebo
Statistical Analysis 2: Comparison: Semaglutide vs Placebo; Analysis for non-fatal myocardial infarction was done by Cox proportional hazards model with treatment (semaglutide; placebo) as a fixed factor and stratified by all possible combinations of the three stratification factors used in the randomisation procedure (in total 9 levels); Test type: Superiority or Other; p = 0.1194, Regression, Cox; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.51 to 1.08] — Semaglutide/Placebo
Statistical Analysis 3: Comparison: Semaglutide vs Placebo; Analysis for non-fatal stroke was done by Cox proportional hazards model with treatment (semaglutide; placebo) as a fixed factor and stratified by all possible combinations of the three stratification factors used in the randomisation procedure (in total 9 levels); Test type: Superiority or Other; p = 0.0438, Regression, Cox; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.38 to 0.99] — Semaglutide/Placebo
Statistical Analysis 4: Comparison: Semaglutide vs Placebo; Analysis for revascularisation was done by Cox proportional hazards model with treatment (semaglutide; placebo) as a fixed factor and stratified by all possible combinations of the three stratification factors used in the randomisation procedure (in total 9 levels); Test type: Superiority or Other; p = 0.0027, Regression, Cox; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.50 to 0.86] — Semaglutide/Placebo
Statistical Analysis 5: Comparison: Semaglutide vs Placebo; Analysis for 'unstable angina requiring hospitalisation' was done by Cox proportional hazards model with treatment (semaglutide; placebo) as a fixed factor and stratified by all possible combinations of the three stratification factors used in the randomisation procedure (in total 9 levels); Test type: Superiority or Other; p = 0.4914, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.47 to 1.44] — Semaglutide/Placebo
Statistical Analysis 6: Comparison: Semaglutide vs Placebo; Analysis for hospitalisation for heart failure was done by Cox proportional hazards model with treatment (semaglutide; placebo) as a fixed factor and stratified by all possible combinations of the three stratification factors used in the randomisation procedure (in total 9 levels); Test type: Superiority or Other; p = 0.5735, Regression, Cox; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.77 to 1.61] — Semaglutide/Placcbo

4. Secondary Outcome: Time From Randomisation to First Occurrence of All-cause Death, Non-fatal MI, or Non-fatal Stroke
Description: Percentage of subjects experiencing a first occurrence of all-cause death, non-fatal MI, or non-fatal stroke.
Time Frame: Time from randomisation up to end of follow-up (scheduled at week 109)
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Semaglutide | Placebo
Number analyzed (Participants) | 1648 | 1649
percentage of subjects | 7.4 | 9.6
Statistical Analysis 1: Comparison: Semaglutide vs Placebo; Analysis for all-cause death, non-fatal MI or non-fatal stroke was done by Cox proportional hazards model with treatment (semaglutide; placebo) as a fixed factor and stratified by all possible combinations of the three stratification factors used in the randomisation procedure (in total 9 levels); Test type: Superiority or Other; p = 0.0292, Regression, Cox; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.61 to 0.97] — Semaglutide/Placebo

5. Secondary Outcome: Change From Baseline to Last Assessment in the Trial in Other Treatment Outcomes: Glycosylated Haemoglobin (HbA1c)
Description: Estimated mean change from baseline in glycosylated haemoglobin (HbA1c) to last assessment in the trial during the treatment period.
Time Frame: Week 0, up to week 104
Population: Full analysis set included all the randomised subjects
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
percentage of glycosylated haemoglobin | -1.09 (0.05) | -1.41 (0.05) | -0.44 (0.05) | -0.36 (0.05)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -0.66, 95% CI 2-sided [-0.80 to -0.52] — Sema 0.5 mg - Placebo 0.5 mg
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.05, 95% CI 2-sided [-1.19 to -0.91] — Sema 1.0 mg - Placebo 1.0 mg

6. Secondary Outcome: Change From Baseline to Last Assessment in the Trial in Other Treatment Outcomes: Fasting Plasma Glucose
Description: Estimated mean change from baseline to last assessment in fasting plasma glucose in the trial during the treatment period.
Time Frame: Week 0, up to week 104
Population: Full analysis set included all the randomised subjects.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
mmol/L | -1.75 (0.12) | -2.11 (0.12) | -1.02 (0.12) | -0.88 (0.12)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -0.72, 95% CI 2-sided [-1.06 to -0.38] — Sema 0.5 mg - Placebo 0.5 mg
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -1.22, 95% CI 2-sided [-1.56 to -0.88] — Sema 1.0 mg - Placebo 1.0 mg

7. Secondary Outcome: Change From Baseline to Last Assessment in the Trial in Other Treatment Outcomes: Body Weight
Description: Estimated mean change from baseline to last assessment in body weight in the trial during the treatment period.
Time Frame: Week 0, up to week 104
Population: Full analysis set included all the randomised subjects. As specified in the protocol, the two placebo dose arms (placebo 0.5 mg + placebo 1.0 mg) were pooled for the analysis of this endpoint.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo
Number analyzed (Participants) | 826 | 822 | 1649
kg | -3.57 (0.21) | -4.88 (0.22) | -0.62 (0.15)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -2.95, 95% CI 2-sided [-3.47 to -2.44] — Sema 0.5 mg - Placebo
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = -4.27, 95% CI 2-sided [-4.78 to -3.75] — Semaglutide 1.0 mg - Placebo

8. Secondary Outcome: Change From Baseline to Last Assessment in the Trial in Other Treatment Outcomes: Lipid Profile
Description: Estimated ratio to baseline at week 104 during the treatment period in lipid profile (total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides).
Time Frame: Week 0, up to week 104
Population: Full analysis set included all randomised subjects.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
mg/dL
  Total cholesterol (mg/dL) | 0.97 (0.01) | 0.97 (0.01) | 1.00 (0.01) | 0.99 (0.01)
  HDL-cholesterol (mg/dL) | 0.99 (0.01) | 1.01 (0.01) | 0.99 (0.01) | 0.97 (0.01)
  LDL-cholesterol (mg/dL) | 0.97 (0.01) | 0.98 (0.01) | 1.01 (0.01) | 0.99 (0.01)
  Triglycerides (mg/dL) | 0.93 (0.01) | 0.92 (0.01) | 0.96 (0.01) | 0.98 (0.01)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for total cholesterol was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit. The response and its baseline value were log-transformed before analysis; Test type: Superiority or Other; p = 0.0149, Mixed Models Analysis; Treatment ratio = 0.97, 95% CI 2-sided [0.95 to 1.00] — Semaglutide 0.5 mg/Placebo 0.5 mg
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.2580, Mixed Models Analysis; Treatment ratio = 0.99, 95% CI 2-sided [0.97 to 1.01] — Semaglutide 1.0 mg/Placebo 1.0 mg
Statistical Analysis 3: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for HDL-cholesterol was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.8106, Mixed Models Analysis; Treatment ratio = 1.00, 95% CI 2-sided [0.99 to 1.02] — Semaglutide 0.5 mg/Placebo 0.5 mg
Statistical Analysis 4: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment ratio = 1.04, 95% CI 2-sided [1.02 to 1.06] — Semaglutide 1.0 mg/Placebo 1.0 mg
Statistical Analysis 5: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for LDL-cholesterol was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.0185, Mixed Models Analysis; Treatment ratio = 0.96, 95% CI 2-sided [0.93 to 0.99] — Semaglutide 0.5 mg/Placebo 0.5 mg
Statistical Analysis 6: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; p = 0.5996, Mixed Models Analysis; Treatment ratio = 0.99, 95% CI 2-sided [0.96 to 1.03] — Semaglutide 1.0 mg/Placebo 1.0 mg
Statistical Analysis 7: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for triglycerides was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.1833, Mixed Models Analysis; Treatment ratio = 0.97, 95% CI 2-sided [0.93 to 1.01] — Semaglutide 0.5 mg/Placebo 0.5 mg
Statistical Analysis 8: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; Treatment ratio = 0.93, 95% CI 2-sided [0.89 to 0.97] — Semaglutide 1.0 mg/Placebo 1.0 mg

9. Secondary Outcome: Change From Baseline to Last Assessment in the Trial in Other Treatment Outcomes: Urinary Albumin to Creatinine Ratio
Description: Estimated ratio to baseline in urinary albumin to creatinine ratio at week 104 during the treatment period.
Time Frame: Week 0, up to week 104
Population: Full analysis set included all the randomised subjects
Measure: Least Squares Mean (Standard Error); unit: mg/g
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
mg/g | 1.02 (0.05) | 0.91 (0.05) | 1.32 (0.07) | 1.29 (0.06)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for urinary albumin to creatinine ration was donne using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit. The response and its baseline value were log-transformed before analysis; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Treatment ratio = 0.78, 95% CI 2-sided [0.68 to 0.89] — Sema 0.5 mg / Placebo 0.5 mg
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; Analysis for urinary albumin to creatinine ration was donne using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment ratio = 0.71, 95% CI 2-sided [0.62 to 0.81] — Sema 1.0 mg / Placebo 1.0 mg

10. Secondary Outcome: Change From Baseline to Last Assessment in the Trial in Other Treatment Outcomes: Vital Signs
Description: Estimated mean change from baseline to last assessment in the trial during the treatment period in vital signs (diastolic blood pressure and systolic blood pressure).
Time Frame: Week 0, up to week 104
Population: Full analysis set included all the randomised subjects.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
mmHg
  Diastolic blood pressure (mmHg) | -1.37 (0.32) | -1.57 (0.32) | -1.42 (0.32) | -1.71 (0.32)
  Systolic blood pressure (mmHg) | -3.44 (0.54) | -5.37 (0.54) | -2.17 (0.54) | -2.78 (0.54)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for diastolic blood pressure was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.9205, Mixed Models Analysis; Treatment difference = 0.04, 95% CI 2-sided [-0.83 to 0.92] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.7477, Mixed Models Analysis; Treatment difference = 0.14, 95% CI 2-sided [-0.74 to 1.03] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 3: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for systolic blood pressure was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.0976, Mixed Models Analysis; Treatment difference = -1.27, 95% CI 2-sided [-2.77 to 0.23] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 4: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Treatment difference = -2.59, 95% CI 2-sided [-4.09 to -1.08] — Semaglutide 1.0 mg - Placebo 1.0 mg

11. Secondary Outcome: Incidence During the Trial in Other Treatment Outcomes: Hypoglycaemic Events
Description: Rates (event rate per 100 exposure years) of severe or blood glucose confirmed symptomatic hypoglycaemia defned as an episode that was severe according to the American diabetic association (ADA) classification or blood glucose (BG) confirmed by a PG value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 0 - 109
Population: Full analysis set included all randomised subjects.
Measure: Number; unit: Event rate per 100 exposure years
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
Event rate per 100 exposure years | 37.5 | 36.2 | 35.3 | 39.7

12. Secondary Outcome: Incidence During the Trial in Other Treatment Outcomes: Adverse Events
Description: Rates (event rate per 100 years of exposure) of treatment emergent adverse events.
Time Frame: Weeks 0-109
Population: Full analysis set included all randomised subjects.
Measure: Number; unit: Event rate per 100 years of exposure
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
Event rate per 100 years of exposure | 330.5 | 337.0 | 317.4 | 298.3

13. Secondary Outcome: Occurrence During the Trial in Other Treatment Outcomes: Anti-semaglutide Antibodies
Description: The percentage of subjects that tested positive for anti-semaglutide antibodies at any time point post-baseline during the trial, from week 0 to week 109.
Time Frame: Weeks 0-109
Population: Full analysis set included all randomised subjects
Measure: Number; unit: Percentage of subjects
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg
Number analyzed (Participants) | 826 | 822
Percentage of subjects | 1.4 | 2.3

14. Secondary Outcome: Change From Baseline to Last Assessment in the Trial in Other Treatment Outcomes: Patient Reported Outcome (PRO)
Description: Estimated mean change from baseline to last assessment in the trial in patient reported outcomes (PRO). PRO questionnaire (SF-36v2TM) measured the individual overall health related quality of life namely bodily pain, general health, mental component summary, mental health, physical component summary, physical functioning, role-emotional, role-physical, social functioning and vitality. The PRO scores were transformed to a 0-100 scale with higher scores indicating greater health related quality of life.
Time Frame: Week 0, up to week 104
Population: Full analysis set included all randomised subjects.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
Scores on a scale
  Bodily pain | 0.66 (0.35) | 1.82 (0.35) | 0.16 (0.35) | 0.35 (0.35)
  General health | 1.66 (0.29) | 2.55 (0.29) | 0.78 (0.29) | 1.13 (0.30)
  Mental component summary | 0.0 (0.35) | 0.86 (0.35) | -0.17 (0.35) | -0.11 (0.35)
  Mental health | 0.48 (0.33) | 1.08 (0.33) | -0.14 (0.33) | -0.31 (0.33)
  Physical component summary | 0.76 (0.28) | 1.74 (0.28) | 0.07 (0.28) | 0.35 (0.28)
  Physical functioning | 0.42 (0.32) | 1.12 (0.32) | -0.38 (0.32) | -0.37 (0.33)
  Role-emotional | 0.17 (0.42) | 0.89 (0.42) | -0.36 (0.42) | -0.05 (0.42)
  Role-physical | 0.39 (0.34) | 1.18 (0.35) | -0.33 (0.35) | 0.03 (0.35)
  Social functioning | -0.25 (0.35) | 0.97 (0.35) | -0.20 (0.36) | -0.17 (0.36)
  Vitality | 0.29 (0.31) | 1.55 (0.31) | -0.04 (0.31) | 0.35 (0.31)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for bodily pain was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.3171, Mixed Models Analysis; Treatment difference = 0.50, 95% CI 2-sided [-0.48 to 1.47] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.0031, Mixed Models Analysis; Treatment difference = 1.47, 95% CI 2-sided [0.50 to 2.45] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 3: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for general health was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.0350, Mixed Models Analysis; Treatment difference = 0.87, 95% CI 2-sided [0.06 to 1.69] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 4: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 3]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Treatment difference = 1.42, 95% CI 2-sided [0.60 to 2.24] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 5: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for mental component summary was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.7277, Mixed Models Analysis; Treatment difference = 0.17, 95% CI 2-sided [-0.79 to 1.13] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 6: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 5]; Test type: Superiority or Other; p = 0.0489, Mixed Models Analysis; Treatment difference = 0.97, 95% CI 2-sided [0.00 to 1.94] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 7: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for mental health was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.1860, Mixed Models Analysis; Treatment Difference = 0.61, 95% CI 2-sided [-0.30 to 1.53] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 8: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis; Treatment difference = 1.39, 95% CI 2-sided [0.48 to 2.31] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 9: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for physical component summary was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.0833, Mixed Models Analysis; Treatment difference = 0.68, 95% CI 2-sided [-0.09 to 1.45] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 10: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 9]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Treatment difference = 1.40, 95% CI 2-sided [0.62 to 2.17] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 11: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for physical functioning was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.0799, Mixed Models Analysis; Treatment difference = 0.80, 95% CI 2-sided [-0.10 to 1.69] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 12: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 11]; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Treatment difference = 1.50, 95% CI 2-sided [0.60 to 2.40] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 13: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for role emotional was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.3717, Mixed Models Analysis; Treatment difference = 0.53, 95% CI 2-sided [-0.63 to 1.68] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 14: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 13]; Test type: Superiority or Other; p = 0.1136, Mixed Models Analysis; Treatment difference = 0.94, 95% CI 2-sided [-0.22 to 2.10] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 15: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for role physical was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.1431, Mixed Models Analysis; Treatment difference = 0.72, 95% CI 2-sided [-0.24 to 1.67] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 16: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 15]; Test type: Superiority or Other; p = 0.0197, Mixed Models Analysis; Treatment difference = 1.14, 95% CI 2-sided [0.18 to 2.11] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 17: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for social functioning was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.9223, Mixed Models Analysis; Treatment difference = -0.05, 95% CI 2-sided [-1.03 to 0.93] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 18: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 17]; Test type: Superiority or Other; p = 0.0237, Mixed Models Analysis; Treatment difference = 1.14, 95% CI 2-sided [0.15 to 2.13] — Semaglutide 1.0 mg - Placebo 1.0 mg
Statistical Analysis 19: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for vitality was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.4523, Mixed Models Analysis; Treatment difference = 0.33, 95% CI 2-sided [-0.53 to 1.19] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 20: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 14, analysis 19]; Test type: Superiority or Other; p = 0.0064, Mixed Models Analysis; Treatment difference = 1.20, 95% CI 2-sided [0.34 to 2.07] — Semaglutide 1.0 mg - Placebo 1.0 mg

15. Secondary Outcome: Change From Baseline to Last Assessment in the Trial in Other Treatment Outcomes: Lipid Profile (Free Fatty Acids)
Description: Estimated ratio to baseline at week 104 during the treatment period in lipid profile (free fatty acids).
Time Frame: Week 0, up to week 104
Population: Full analysis set included all randomised subjects.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
mmol/L | 0.95 (0.02) | 0.91 (0.01) | 0.96 (0.02) | 0.99 (0.02)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for free fatty acids was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p = 0.7796, Mixed Models Analysis; Treatment ratio = 0.99, 95% CI 2-sided [0.95 to 1.04] — Semaglutide 0.5 mg/Placebo 0.5 mg
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Treatment ratio = 0.92, 95% CI 2-sided [0.88 to 0.96] — Semaglutide 1.0 mg/Placebo 1.0 mg

16. Secondary Outcome: Change From Baseline to Last Assessment in the Trial in Other Treatment Outcomes: Vital Signs (Pulse Rate)
Description: Estimated mean change from baseline to last assessment in the trial during the treatment period in vital signs (pulse rate).
Time Frame: Week 0, up to week 104
Population: Full analysis set included all the randomised subjects.
Measure: Least Squares Mean (Standard Error); unit: beats/min
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Number analyzed (Participants) | 826 | 822 | 824 | 825
beats/min | 2.12 (0.34) | 2.41 (0.34) | 0.09 (0.34) | -0.07 (0.34)
Statistical Analysis 1: Comparison: Semaglutide 0.5 mg vs Placebo 0.5 mg; Analysis for pulse rate was done using a mixed model for repeated measurements with treatment (4 levels) and stratification (9 levels) as fixed factors and baseline value as covariate, all nested within visit; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = 2.02, 95% CI 2-sided [1.07 to 2.98] — Semaglutide 0.5 mg - Placebo 0.5 mg
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Placebo 1.0 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment difference = 2.47, 95% CI 2-sided [1.52 to 3.43] — Semaglutide 1.0 mg - Placebo 1.0 mg

ADVERSE EVENTS:
Time Frame: Adverse events from the first trial-related activity after the subject had signed the informed consent (week -2) until the end of the posttreatment follow-up period (week 109).
Description: Safety was assessed using the full analysis set which included all randomised subjects. Subjects contributed to the evaluation as randomised.
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Placebo 0.5 mg | Placebo 1.0 mg
Serious Adverse Events (participants affected / at risk) | 289/826 | 276/822 | 329/824 | 298/825
Other Adverse Events (participants affected / at risk) | 573/826 | 587/822 | 547/824 | 524/825
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=826) | Semaglutide 1.0 mg (N=822) | Placebo 0.5 mg (N=824) | Placebo 1.0 mg (N=825)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (3) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Accident at work (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 4 (4) | 3 (3) | 1 (1) | 2 (2)
Acute hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 18 (22) | 6 (8) | 14 (14) | 22 (24)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 16 (21) | 13 (14) | 15 (15) | 27 (28)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 4 (4) | 2 (2) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 9 (9) | 9 (10) | 16 (17) | 12 (12)
Angina unstable (Cardiac disorders) | 13 (16) | 15 (18) | 19 (21) | 22 (23)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (2) | 1 (1) | 1 (1) | 3 (3)
Arterial insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriogram coronary (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 14 (16) | 12 (15) | 20 (22) | 18 (19)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 6 (6)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder trabeculation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blindness (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose fluctuation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (6) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Boutonneuse fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brachytherapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bundle branch block left (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 5 (6) | 2 (2) | 3 (3) | 2 (3)
Cardiac asthma (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 10 (11) | 10 (10) | 7 (9) | 3 (4)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 8 (8) | 4 (4) | 6 (6) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 21 (31) | 14 (17) | 15 (19) | 18 (21)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Carotid artery stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Carotid revascularisation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (6)
Cataract cortical (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Catheterisation cardiac (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 6 (6) | 3 (3) | 7 (7) | 9 (10)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 2 (3) | 3 (3) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 3 (3) | 6 (6) | 6 (8)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 3 (3) | 5 (6) | 3 (3)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 0 (0) | 6 (6) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 4 (4) | 2 (2) | 4 (4) | 1 (1)
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chondrolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 10 (10) | 5 (5) | 14 (17) | 5 (5)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 5 (5) | 7 (7) | 7 (9)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 1 (1) | 4 (4) | 5 (5)
Coronary arterial stent insertion (Surgical and medical procedures) | 15 (19) | 8 (9) | 17 (18) | 17 (19)
Coronary artery bypass (Surgical and medical procedures) | 8 (8) | 5 (5) | 14 (14) | 10 (10)
Coronary artery disease (Cardiac disorders) | 11 (11) | 9 (9) | 5 (6) | 2 (3)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 7 (7) | 2 (2) | 4 (4) | 1 (1)
Coronary revascularisation (Surgical and medical procedures) | 11 (12) | 10 (10) | 15 (17) | 9 (10)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystoid macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 5 (7) | 4 (5)
Diabetic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 6 (8) | 2 (2) | 3 (3) | 5 (8)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Diabetic mononeuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 4 (4) | 2 (3) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dural tear (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 3 (3) | 4 (4)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram ST segment abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epididymal tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eyelid dermatochalasis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to anastomose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 11 (11) | 5 (5) | 11 (11) | 8 (8)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder necrosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 4 (4) | 2 (2)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (1) | 4 (4)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Glomerulonephritis chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Growth hormone-producing pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic congestion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 4 (4) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Hypertensive emergency (Vascular disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia malignant (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (8) | 2 (2) | 5 (7) | 6 (6)
Hypoglycaemic unconsciousness (Nervous system disorders) | 5 (5) | 3 (3) | 1 (1) | 3 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intra-abdominal haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 8 (8) | 7 (8) | 16 (16) | 4 (4)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laparotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mechanical ventilation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Metaplasia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Microlithiasis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Movement disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 4 (5) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4) | 10 (10) | 9 (10) | 12 (14)
Myocardial ischaemia (Cardiac disorders) | 6 (6) | 2 (2) | 3 (3) | 2 (2)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 8 (8) | 5 (5) | 8 (8) | 4 (5)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (8) | 9 (9) | 10 (10)
Osteomyelitis (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 3 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otosclerosis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic enzymes increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Parkinsonism (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 2 (2) | 1 (1) | 3 (4) | 6 (7)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery angioplasty (Surgical and medical procedures) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Peripheral artery bypass (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral artery stent insertion (Surgical and medical procedures) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Peripheral endarterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral revascularisation (Surgical and medical procedures) | 2 (2) | 4 (4) | 5 (5) | 9 (9)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Periumbilical abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 18 (19) | 15 (16) | 22 (26) | 14 (14)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Post procedural pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Proctitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3) | 4 (4) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Pterygium operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 3 (3) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (6)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Radiculitis lumbosacral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Removal of internal fixation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal artery arteriosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 3 (3) | 3 (3)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Retinopathy haemorrhagic (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 3 (3) | 4 (5)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 7 (7) | 4 (4) | 3 (3) | 7 (7)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (2)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep terror (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Splenic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Stent placement (Surgical and medical procedures) | 2 (2) | 2 (2) | 1 (1) | 1 (2)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 4 (4) | 3 (4) | 3 (3)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 7 (8) | 6 (7) | 10 (10) | 7 (7)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (9) | 2 (2) | 10 (10) | 6 (6)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
VIth nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular asystole (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Ventricular hypokinesia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 8 (8) | 1 (2) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Volvulus of small bowel (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspergilloma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cor pulmonale acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic end stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leriche syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumobilia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal artery stent placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic encephalopathy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon sheath incision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=826) | Semaglutide 1.0 mg (N=822) | Placebo 0.5 mg (N=824) | Placebo 1.0 mg (N=825)
Abdominal pain (Gastrointestinal disorders) | 45 (54) | 35 (40) | 33 (37) | 31 (36)
Abdominal pain upper (Gastrointestinal disorders) | 35 (37) | 42 (53) | 19 (22) | 19 (33)
Amylase increased (Investigations) | 31 (39) | 48 (57) | 28 (33) | 28 (33)
Anaemia (Blood and lymphatic system disorders) | 41 (46) | 33 (34) | 44 (46) | 48 (55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 (45) | 35 (40) | 57 (69) | 58 (70)
Back pain (Musculoskeletal and connective tissue disorders) | 54 (54) | 49 (58) | 49 (59) | 48 (50)
Bronchitis (Infections and infestations) | 46 (52) | 38 (43) | 49 (52) | 51 (64)
Cataract (Eye disorders) | 55 (59) | 43 (48) | 37 (38) | 45 (46)
Constipation (Gastrointestinal disorders) | 46 (52) | 79 (97) | 37 (42) | 36 (38)
Decreased appetite (Metabolism and nutrition disorders) | 86 (97) | 75 (88) | 19 (21) | 9 (10)
Diabetic retinopathy (Eye disorders) | 46 (50) | 56 (63) | 39 (39) | 38 (43)
Diarrhoea (Gastrointestinal disorders) | 148 (277) | 148 (245) | 97 (159) | 87 (112)
Dizziness (Nervous system disorders) | 53 (57) | 46 (54) | 38 (53) | 38 (45)
Dyspepsia (Gastrointestinal disorders) | 51 (68) | 63 (88) | 23 (25) | 18 (19)
Headache (Nervous system disorders) | 54 (77) | 58 (89) | 67 (114) | 74 (110)
Influenza (Infections and infestations) | 51 (60) | 48 (56) | 48 (57) | 46 (63)
Lipase increased (Investigations) | 94 (121) | 90 (123) | 66 (76) | 69 (83)
Nasopharyngitis (Infections and infestations) | 66 (91) | 60 (77) | 78 (99) | 66 (84)
Nausea (Gastrointestinal disorders) | 143 (233) | 179 (282) | 62 (78) | 66 (94)
Upper respiratory tract infection (Infections and infestations) | 53 (59) | 51 (64) | 63 (75) | 65 (88)
Urinary tract infection (Infections and infestations) | 78 (108) | 71 (93) | 64 (97) | 68 (87)
Vomiting (Gastrointestinal disorders) | 87 (128) | 122 (170) | 42 (51) | 33 (41)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (41) | 32 (33) | 40 (41) | 46 (48)
Fatigue (General disorders) | 24 (27) | 42 (48) | 15 (16) | 26 (28)
Microalbuminuria (Renal and urinary disorders) | 27 (30) | 33 (35) | 46 (51) | 42 (45)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 (42) | 29 (31) | 46 (51) | 42 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.